CLINICAL TRIAL: NCT01750463
Title: Verifying the Accuracy of the Masimo Pronto Non-Invasive Hemoglobin (Hb) Monitor and Associated Rainbow Probes Compared to Measured Laboratory Values in Critically Ill Pediatric Patients
Brief Title: Comparing Validity of Non-Invasive Hemoglobin Monitoring to Laboratory Results in Critically Ill Children
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Sean McLean, MD, MD, University of North Carolina, Chapel Hill
Other Study IDs: 12-2019
Record Dates: First submitted 2012-12-05; First posted 2012-12-17 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Hemoglobin Results
Keywords: Pediatric critically ill; Masimo; hemoglobin; monitoring; UNC; PICU

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm A: Critically ill pediatric patients admitted to PICU requiring hemoglobin monitoring.
  Patients admitted to PICU requiring hemoglobin monitoring will have a reading total hemoglobin (SpHb) assessment done with the Masimo Pronto Rad 7 Non-Invasive hemoglobin monitor,prior to standard laboratory blood draw and hemoglobin analysis.
  Interventions: Other: Masimo Pronto Rad 7 Non-Invasive hemoglobin monitor; Other: Standard Laboratory Blood Draw and Hemoglobin Analysis

INTERVENTIONS:
Other: Masimo Pronto Rad 7 Non-Invasive hemoglobin monitor — Patients admitted to PICU requiring hemoglobin monitoring will have a total hemoglobin (SpHb) assessment from Masimo non-invasive monitor, prior to standard, required blood draw and laboratory analysis.
  Other Names: Rainbow adhesive sonsor R1 20L; Rainbow reusable spot check sensor DCIP SC-200; Rainbow reusable spot check sensor DCI SC-200
Other: Standard Laboratory Blood Draw and Hemoglobin Analysis — Patients admitted to PICU requiring hemoglobin monitoring will have a reading from Masimo non-invasive monitor, prior to standard, required blood draw and laboratory analysis.

SUMMARY:
This is a prospective study to determine the accuracy of the Masimo Pronto Non-Invasive Hemoglobin Monitor and associated Rainbow® probes in the detection of hemoglobin concentration in critically ill children.

DETAILED DESCRIPTION:
This is a prospective study to determine the accuracy of the Masimo Pronto Non-Invasive Hemoglobin Monitor and associated Rainbow® probes in the detection of hemoglobin concentration in critically ill children. Data from at least 30 patients admitted to the Pediatric Intensive Care Unit (PICU) over a period of 2 months will be collected and analyzed for this study.

Note, that this device would not lead to deviations in routine patient care; specifically, the non-invasive monitor placed on the patient's finger is FDA approved. The proposed monitors are identical macroscopically to monitors, which are currently used to measure oxygen saturation at this institution. Clinical decisions, additional blood draws or alterations to the plan of care will not be made based on study data. The objective is to compare the validity of the hemoglobin values determined from non-invasive technology with measured laboratory values for hemoglobin utilized as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been admitted to Pediatric Intensive Care Unit
* Patient age is ≥ 30 days old and ≤ 18 years old
* Patient weight ≥ 3 Kg.
* Patient requires hemoglobin monitoring

Exclusion Criteria:

* Patient does not have exposed fingers/toes,due to congenital anomalies wound dressing or injury.
* Patient weight is less than 3 Kg
* Patient is less than 30 days old

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients admitted to the PICU requiring hemoglobin monitoring
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Comparison of standard hemoglobin monitoring vs. the MASIO non-invasive hemoglobin monitor | up to 48 hours, post PICU admission
  We will obtain measurements using the Masimo Pronto device prior to the standard lab draw at the following time points: post admission to PICU, 12-48 hours. We will then perform analysis using Bland Altman methods to determine the degree of agreement.
  Data analysis will occur 1 year after enrollment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Phillips, MD, Principal Investigator — University of North Carolina,Chapel Hill, NC
Locations (1):
- Pediatric Intensive Care Unit, University of North Carolina, Chapel Hill, North Carolina, United States